CLINICAL TRIAL: NCT07400562
Title: Electrophysiological Effects of Adjunct Low-Level Laser Therapy and Median Nerve Mobilization After Carpal Tunnel Release: A Randomized Controlled Study
Brief Title: Electrophysiological Effects of Adjunct Low-Level Laser Therapy and Median Nerve Mobilization After Carpal Tunnel Release
Acronym: LL-CTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galala University (Other)
Responsible Party: Principal Investigator, Eman Hamed, Lecturer of Clinical Pharmacy, Galala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Low-Level Laser Therapy -LLCTR; Galala University (Other: i am faculty of pharmacy galala university-This study was approved by the Ethical Committee of the Faculty of physical)
Record Dates: First submitted 2026-01-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal tunnel syndrome; Neuropathy; Low-level laser therapy; Median nerve mobilization
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — gallium arsenide

STUDY DESIGN:
Intervention Model Description: This study was designed as a prospective, parallel-group, randomized controlled trial. Eligible participants who had undergone unilateral carpal tunnel release were randomly assigned to one of three intervention arms in a 1:1:1 allocation ratio. Group A received adjunct low-level laser therapy, Group B received median nerve mobilization exercises, and Group C received standard postoperative care without adjunctive therapy. Randomization was performed using a concealed allocation method. Outcomes were assessed at baseline and after 6 weeks of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LLLT (GaAs 904-nm Laser) Group (Experimental): - Patients in group (A) had a regimen of infrared Gallium Arsenide low-level laser therapy (20 mW average power, 904 nm wavelength, laser probe diameter of 7 mm). The treatment was administered to the palmar region above the carpal tunnel and along the median nerve pathway, with a cumulative dosage of 4.8 J
  Interventions: Other: Gallium Arsenide (GaAs) 904-nm Low-Level Laser Device
- Median Nerve Mobilization Group (Experimental): Patients in the group (B) were instructed to do a series of movements that included the median nerve: lateral rotation of the shoulders, depression, wrist extension, supination, shoulder abduction, elbow extension, and bending the neck laterally to the other side.
  Interventions: Other: Therapist-Supervised Median Nerve Neural Mobilization Exercises
- Standard Care Control Group (Experimental): Control group
  Interventions: Other: Standard Postoperative Care

INTERVENTIONS:
Other: Gallium Arsenide (GaAs) 904-nm Low-Level Laser Device — Group A: GaAs diode laser, 904 nm, average power 20 mW, probe diameter 7 mm (spot size approximately 0.385 cm²), administered as 1.2 J per point at four standardized points (totaling 4.8 J per session); 60 seconds per point (totaling approximately 4 minutes per session). Over 18 sessions (3 per week for 6 weeks), the total energy administered per treatment cycle is 86.4 J. This methodology and point-based dosing method were chosen to align with prevalent CTS protocols utilizing identical device specifications and total-session dosage, while adhering to the required 904-nm dosing parameters
  Arms: LLLT (GaAs 904-nm Laser) Group
Other: Therapist-Supervised Median Nerve Neural Mobilization Exercises — Patients in the group (B) were instructed to do a series of movements that included the median nerve: lateral rotation of the shoulders, depression, wrist extension, supination, shoulder abduction, elbow extension, and bending the neck laterally to the other side. They were directed to maintain the final posture for 20 seconds. Therapist-supervised median nerve mobilization was performed three sessions/week for 6 weeks; each session included three sets of 5 repetitions of the standardized sequence, with the end-position held for 20 seconds per repetition and ~10 seconds rest between repetitions (and ~60 seconds rest between sets). Total mobilization time was ~10-12 minutes per session, and all sessions were conducted under direct therapist supervision to ensure correct positioning and symptom monitoring
  Arms: Median Nerve Mobilization Group
Other: Standard Postoperative Care — Group C patients served as the comparison (control) group.
  Arms: Standard Care Control Group

SUMMARY:
This randomized controlled study investigated whether adding low-level laser therapy (LLLT) or median nerve mobilization after unilateral carpal tunnel release improves median nerve electrophysiological parameters compared with no adjunctive treatment. Forty-five patients were randomly assigned to receive LLLT, median nerve mobilization, or standard postoperative care. Interventions were delivered over six weeks, and nerve conduction studies were conducted before and after treatment to assess electrophysiological outcomes, with motor distal latency designated as the primary outcome measure.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is commonly managed surgically through carpal tunnel release (CTR); however, postoperative recovery may be accompanied by persistent neural dysfunction and delayed nerve conduction improvement. Adjunct rehabilitation strategies, such as low-level laser therapy (LLLT) and median nerve mobilization, have been proposed to enhance neural recovery, yet their electrophysiological effects following CTR remain insufficiently established.

This randomized controlled study aimed to examine and compare the effects of adjunct LLLT and median nerve mobilization on median nerve electrophysiological parameters after unilateral CTR. Forty-five patients diagnosed with unilateral CTS and treated surgically with CTR were recruited. Participants (aged 25-55 years) were randomly allocated into three equal groups. Group A received adjunct gallium arsenide (GaAs) infrared LLLT, Group B underwent median nerve mobilization exercises, and Group C received standard postoperative care without adjunctive therapy.

Both intervention protocols were applied three times per week for six consecutive weeks. Electrophysiological assessments were conducted at baseline (pre-intervention) and after six weeks using standardized nerve conduction studies. Measured parameters included motor distal latency (MDL), sensory distal latency (SDL), motor nerve conduction velocity (MCV), and compound motor action potential amplitude (CMAP), with MDL predefined as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

Age between 25 and 55 years Clinical diagnosis of unilateral carpal tunnel syndrome Underwent surgical carpal tunnel release (transverse carpal ligament release)

Exclusion Criteria:

Rheumatoid arthritis Diabetes mellitus History of wrist fracture or other wrist joint trauma Current use of anti-inflammatory medications or other interfering medications Receipt of alternative treatments (e.g., acupuncture, physical therapy modalities) Use of wrist orthoses

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Change in Median Nerve Motor Distal Latency | 6 weeks
  Change in motor distal latency (milliseconds) of the median nerve from baseline (pre-treatment) to 6 weeks post-intervention, assessed using standardized nerve conduction testing (Neuropack) following American Association of Electrodiagnostic Medicine guidelines.

SECONDARY OUTCOMES:
Change in Median Nerve Sensory Distal Latency | 6 weeks
  Change in sensory distal latency (milliseconds) of the median nerve from baseline to 6 weeks post-intervention.
Change in Median Nerve Motor Conduction Velocity | 6 weeks
  Change in motor nerve conduction velocity (meters/second) of the median nerve from baseline to 6 weeks post-intervention.
Change in Compound Motor Action Potential Amplitude | 6 weeks
  Change in CMAP amplitude (millivolts) of the median nerve from baseline to 6 weeks post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Giza Governorate, Egypt